CLINICAL TRIAL: NCT01783951
Title: Autologous Dendritic Cell-cytokine Induced Killer Cell Immunotherapy Combined With S-1 Based Chemotherapy in Patients With Advanced Gastric Cancer
Brief Title: Study of S-1 Plus DC-CIK for Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Duke University (Other); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director,Capital Medical University (CMU)Cancer Center, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1+DC CIK- G
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; S-1; DC-CIK; T cell
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC-CIK plus S-1 based chemotherapy (Experimental): Patients will be receive S-1 based chemotherapy, including S-1 plus cisplatin or S-1 alone. Meanwhile those patients will receive DC-CIK cell therapy at days 15, 17 and 19 per cycle and received cycles of treatment once every 21 days.Treatment was continued until disease progression, unacceptable toxic effects, or the withdrawal of consent.
  Interventions: Biological: DC-CIK; Drug: S-1; Drug: Cisplatin
- S-1 based chemotherapy (Active Comparator): Patients will be receive S-1 based chemotherapy, including S-1 plus cisplatin or S-1 alone.Cycles were repeated every 21 days. Treatment was continued until disease progression, unacceptable toxic effects, or the withdrawal of consent.
  Interventions: Drug: S-1; Drug: Cisplatin

INTERVENTIONS:
Biological: DC-CIK — Patients will be receive DC-CIK cell therapy at days 15, 17 and 19 per cycle and received cycles of treatment once every 21 days.
  Arms: DC-CIK plus S-1 based chemotherapy
Drug: S-1 — The dose of S-1 is determined according to the body surface area as follows: <1.25 m2, 40 mg; 1.25 to <1.5 m2, 50 mg; and ≥1.5 m2, 60 mg, given twice daily after meals for 14 days followed by 7 days rest.
Drug: Cisplatin — Cisplatin is administered at 75 mg/m2 intravenously over 1 to 3 hours every 21 days.

SUMMARY:
The purpose of this study is to evaluate the antitumor effect and safety of clinical effectiveness dendritic cell activated Cytokine induced killer treatment (DC-CIK) plus S-1 based chemotherapy for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed recurrent or metastatic gastric or esophagogastric junctional adenocarcinoma
* Between 18 and 80 years old
* Capable of oral intake
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Karnofsky Performance Status (KPS) ≥ 70%
* Normal functions of heart, lung and bone marrow
* Adequate hematological profile： Hemoglobin ≥ 9.0 g/dL Absolute granulocyte count ≥ 1,500/mm3 Platelet count ≥ 100,000/mm3
* Adequate hepatic function Total bilirubin level≤ 3.0 times the upper limit of normal (ULN) Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN
* Adequate renal function(normal serum creatinine level)
* A life expectancy≥ 2 months
* Informed consent signed

Exclusion Criteria:

* Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study
* Any radiotherapy or surgery within the previous 4 weeks
* Symptomatic brain metastasis not controlled by corticosteroids
* Bone marrow metastasis
* Active infection
* Serious complications
* Receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1: phenytoin, potassium warfarin , flucytosine, cimetidine and folinic acid.
* Pregnant or lactation women, or women with known or suspected pregnancy and men who want let to pregnancy
* Ineligible for the study at the discretion of investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival（PFS） | 4 years

SECONDARY OUTCOMES:
Overall survival | 4 years
Response rate | Every 6 weeks
Adverse Events | Every 3 weeks
Quality of life | 6 weeks
  Evaluation of quality of life will be performed every 2 cycles (6 weeks) from baseline to the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Cancer Center, Beijing, Beijing Municipality, China